CLINICAL TRIAL: NCT04850118
Title: A Randomized, Controlled, Masked, Multi-center Study Evaluating the Efficacy, Safety, and Tolerability of Two Doses of AGTC-501 Compared to an Untreated Control Group in Male Participants With X-linked Retinitis Pigmentosa
Brief Title: A Clinical Trial Evaluating the Safety and Efficacy of a Single Subretinal Injection of AGTC-501 in Participants With XLRP
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Beacon Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AGTC-RPGR-002
Record Dates: First submitted 2021-04-05; First posted 2021-04-20 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: X-Linked Retinitis Pigmentosa
Keywords: XLRP; retinal degeneration; RPGR; adeno-associated virus; AAV; gene therapy
MeSH Terms: conditions — Retinal Degeneration

STUDY DESIGN:
Intervention Model Description: Participants are randomized in a 1:1:1 ratio to 1 of 3 groups (high dose, low dose, untreated) control. After 12 months, participants in the untreated group will be evaluated to determine eligibility to receive the high dose of AGTC-501.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For groups 1 and 2 (AGTC-501 dosing groups), both the participants and the Investigators are masked to dose assignment, and only the unmasked staff who prepare the dose are unmasked to the participants dose assignment. Due to the need to perform the subretinal injection to administer the study drug, both participants and Investigators will know whether the participant was assigned to a treatment group or to the control group. To minimize bias of the treated and control study eye evaluations, starting at Month 3, microperimetry, and BCVA/LLVA assessments will be conducted by appropriately qualified masked evaluators who do not know whether the participant underwent surgery. Participants will be instructed not to disclose whether they had surgery to the examiner administering the test.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Group 1: Dose (Active Comparator): Male participants 12-50 years of age treated by subretinal injection with the of AGTC-501
  Interventions: Biological: rAAV2tYF-GRK1-hRPGRco
- Group 2: Dose (Active Comparator): Male participants 12-50 years of age treated by subretinal injection with the dose of AGTC-501
  Interventions: Biological: rAAV2tYF-GRK1-hRPGRco
- Group 3: Control (Other): Male participants 12-50 years of age in the untreated control group. Participants in the control group will be followed for a minimum of 24 months. After all participants have reached Month 12, participants in the control group will be given the option to receive the study drug in the fellow eye, if eligible.
  Interventions: Drug: Control

INTERVENTIONS:
Biological: rAAV2tYF-GRK1-hRPGRco — Adeno-associated virus vector expressing a human RPGR gene
  Other Names: AGTC-501
  Arms: Group 1: Dose; Group 2: Dose
Drug: Control — Untreated Control Group 3
  Other Names: Untreated Control Group
  Arms: Group 3: Control

SUMMARY:
This study will evaluate and compare the safety, efficacy, and tolerability of 2 doses of a recombinant adeno-associated virus vector (AGTC-501/laruparetigene zovaparvovec )) to an untreated control group in male participants with X-linked retinitis pigmentosa caused by RPGR mutations.

DETAILED DESCRIPTION:
This study is a randomized, controlled, masked, multi-center study evaluating and comparing 2 doses of AGTC-501 to an untreated control group. A single subretinal injection of AGTC-501 Dose 1 or Dose 2 will be administered in participants in 2 treatment groups while participants in the untreated control group will be followed and evaluated, after which they will be evaluated to determine eligibility to receive treatment with AGTC-501 Dose 2.

Approximately 75 eligible male participants between 12 and 50 years of age (inclusive) will be randomized in a 1:1:1 ratio to 1 of 3 groups.

ELIGIBILITY:
General Inclusion Criteria:

1. Provide written informed consent or assent (per local regulation), prior to the conduct of any study-related procedure. Participants who provide assent must have a parent, guardian, or legal representative provide written informed consent.
2. Be between 12 and 50 years of age (inclusive) at the time of informed consent and assent (as applicable).
3. Be male (XY chromosome) and have at least one documented pathogenic or likely pathogenic variant in the RPGR gene.
4. Have a clinical diagnosis of XLRP.
5. Be able and willing, as assessed by the Investigator, to follow study instructions, complete study assessments, comply with the protocol, and attend study visits for the duration of the study.

   Ocular Inclusion Criteria (Study Eye):
6. Have a BCVA ≤ 78 letters (approximately Snellen, 20/32) and ≥ 34 letters (approximately Snellen, 20/200)
7. Have a LLVA ≤64 letters (approximately Snellen 20/50) in the study eye
8. Be able to perform all tests of visual and retinal function and structure in both eyes based on the participant's reliability, and fixation, in the study eye per the Investigator's discretion.
9. Have an LLD of > 10 letters in the study eye
10. Have detectable baseline mean macular sensitivity measured by MAIA microperimetry, between 1-12 decibels (dB) in the study eye, as determined by the Investigator and confirmed by the CRC with fixation loss ≤20% at each screening visit.
11. Have a detectable sub-foveal EZ line in the study eye as assessed by spectral domain-optical coherence tomography (SD-OCT) and confirmed by the CRC.

General Exclusion Criteria:

1. Have other known disease-causing mutations documented in the participant's medical history or identified through a retinal dystrophy gene panel, that in the opinion of the Investigator would interfere with the potential therapeutic effect of the study agent or the quality of the assessments.
2. For participants with herpes simplex virus (HSV):

   1. Have history of oral or genital herpes and unable and/or unwilling to utilize prophylactic antiviral medication.
   2. Have a history of ocular herpes.
   3. Have active oral or genital herpes or are currently receiving treatment for HSV infection.
3. Have known sensitivity or allergy to systemic corticosteroids or other immunosuppressive medications.
4. Have used anti-coagulant agents that may alter coagulation
5. Have used systemic corticosteroids or other immunosuppressive medications within 3 months prior to screening and/or intend to use during screening. Corticosteroids used on an as-needed basis administered by insufflation, inhalation or local administration to the skin
6. If sexually active or planning to become sexually active, are unwilling to use barrier contraception for 3 months following treatment administration.
7. Are currently participating or recently participated in any other research
8. Have previously received any AAV gene therapy product, stem cell therapy, cell-based therapy, or similar biologics.
9. Have significant media opacity impacting evaluation of the retina or vitreous. administration.
10. Had intraocular surgery within 90 days of study treatment administration.
11. Have any active ocular/intraocular infection or inflammation
12. Have a history of corticosteroid-induced raised IOP of >25 mmHg following corticosteroid exposure, despite topical IOP-lowering pharmacologic therapy.
13. Have any artificial retinal implant or prosthesis.
14. Have absence of clear ocular media and/or inadequate pupil dilation to facilitate good quality SD-OCT images.
15. Have any history of rhegmatogenous retinal detachment.
16. Have myopia (spherical equivalent) exceeding -10 diopters (or axial length of >30 mm if the Principal Investigator [PI] deems it appropriate to measure) or presence of pathologic myopia in the study eye.
17. Have passed the Low Contrast Ora-VNC mobility course at ≤0.35 lux light level in either eye or binocularly at any screening visit.

Ages: 12 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Enrollment: 85 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
The proportion of participants with a ≥15 letter increase from baseline in LLVA | Day 0 - Month 12
  LLVA(Low Luminance Visual Acuity) will be determined by adding a neutral density filter to the refraction using standard ETDRS (Early Treatment of Diabetic Retinopathy) visual acuity or tumbling "E" chart

SECONDARY OUTCOMES:
Change from baseline in LLVA (First Key Secondary Endpoint) | Day 0 - Month 12
  Functional vision will be determined by adding a neutral density filter to the refraction using standard ETDRS (Early Treatment of Diabetic Retinopathy) visual acuity or tumbling "E" chart
Change from baseline in mean sensitivity across the whole grid, as measured by MAIA (Second Key Secondary Endpoint) microperimetry | Day 0 - Month 12
  As assessed by MAIA (Macular Integrity Assessment) microperimetry - assess photoreceptor function under low-light
Change from baseline in full-field stimulus threshold (FST) (Third Key Secondary Endpoint) | Day 0 - Month 12
  Full-field stimulus threshold (FST) measures the sensitivity of the visual field by testing for the lowest luminance flash which elicits a visual sensation perceived

OTHER OUTCOMES:
Number and proportion of treatment-emergent ocular/non-ocular adverse events | Day 0 - Year 5
  Ocular/non-ocular adverse events are collected the duration of the trial

CONTACTS AND LOCATIONS:
Overall Officials: Carrie Reichley, Study Director — Beacon Therapeutics
Locations (24):
- United States (19):
  - Retina Macula Institute of Arizona, Scottsdale, Arizona
  - Children's Hospital Los Angeles, Los Angeles, California
  - University of Florida Health Jacksonville, Department of Ophthalmology, Jacksonville, Florida
  - Bascom Palmer Eye Institute- University of Miami, Miami, Florida
  - Midwest Eye Institute (Retina Partners Midwest), Carmel, Indiana
  - Wilmer Eye Institute at Johns Hopkins, Baltimore, Maryland
  - Ophthalmic Consultants of Boston, Boston, Massachusetts
  - Mayo Clinic, Rochester, Minnesota
  - Duke Eye Center, Durham, North Carolina
  - Cincinnati Eye Institute, Cincinnati, Ohio
  - Cole Eye Institute - Cleveland Clinic, Cleveland, Ohio
  - Casey Eye Institute, OHSU, Portland, Oregon
  - The Center for Advanced Retinal & Ocular Therapeutics University of Pennsylvania Perelman School of Medicine, Philadelphia, Pennsylvania
  - Mid Atlantic Retina, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Retina Consultants of Texas, Bellaire, Texas
  - Retina Foundation of the Southwest, Dallas, Texas
  - Baylor Eye Institute, Houston, Texas
  - Retina Consultants of San Antonio Texas, San Antonio, Texas
- Australia (2):
  - Sydney Eye Hospital, Sydney, New South Wales
  - Royal Victorian Eye & Ear Hospital, East Melbourne, Victoria
- United Kingdom (3):
  - Moorfields Eye Hospital, London
  - The Retina Clinic London, Institute of Ophthalmology, University College London, London
  - Oxford Eye Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang CY, Chen L, Lin TY, Huang SP. Systematic Identification of Candidate Genes for Inherited Retinal Disease Gene Therapy Integrating Worldwide IRD Cohort and Single-Cell Analysis. J Ophthalmol. 2025 Jun 12;2025:7014745. doi: 10.1155/joph/7014745. eCollection 2025. PMID 40547876